CLINICAL TRIAL: NCT01427452
Title: Kidney Donor Outcomes Cohort (KDOC) Study
Acronym: KDOC
Status: Completed | Type: Observational
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, James Rodrigue, Professor, Beth Israel Deaconess Medical Center
Other Study IDs: 2010P000286; R01DK085185 (NIH)
Record Dates: First submitted 2011-08-30; First posted 2011-09-01 (Estimated); Last update posted 2018-03-20 (Actual); Status verified 2018-03

CONDITIONS: Living Donor Nephrectomy
Keywords: Live Donor; Kidney Donation; Living Donation; Live Donor Kidney Transplantation; Donor Nephrectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Living Kidney Donor, Transplant Recipient, Healthy Control: Living kidney donors and their transplant recipient will be enrolled. Also, a smaller cohort of healthy controls (potential donors who were medically suitable but not used) will be enrolled.

SUMMARY:
Live donor kidney transplantation (LDKT) is important because its outcomes for recipients are superior to those of deceased donor transplantation, and it yields significant cost savings to the healthcare system overall. Despite efforts over the past few decades to enhance understanding of the short- and long-term outcomes of living kidney donation, it is clear that investigators have more knowledge in some areas (e.g., surgical and medical complications) than in others (e.g., psychological outcomes, financial impact). While the transplant community and changes in federal regulations have brought attention to the need for more systematic study of living donor outcomes, there remains a paucity of scientifically rigorous multisite, prospective outcome studies. The long-term goal of this research program is to characterize the short- and long-term surgical, medical, functional, psychological, and financial outcomes of living kidney donation. The objective of this study is to establish a multisite prospective cohort of living kidney donors, their recipients, and a healthy comparison group. This cohort will be used to examine three primary aims: (1) to assess donor outcomes (surgical, medical, functional, psychological, financial) over a 2-year period initially, with the intention of examining these outcomes over a more extended time period in subsequent years; (2) to identify the donor, recipient, and center variables that are most predictive of donor outcomes; and (3) to identify disparities in donor outcomes and their predictors. To accomplish these aims, six kidney transplant programs, representing six states (Massachusetts, Maine, Rhode Island, New York, Iowa, and Arizona) and with experience and expertise in caring for living donors and transplant recipients, will participate in the study. Donors, their recipients, and healthy controls will complete comprehensive assessments at baseline (pre-surgery) and at 1, 6, 12, and 24 months post-donation. This study will extend the investigators considerable preliminary work by simultaneously examining outcomes that are of importance to donors, recipients, healthcare providers, and policymakers. The rationale for this research is that, once these outcomes and their predictors are known, investigators can further develop and refine educational strategies and informed consent processes for both living donors and their intended recipients, as well as provide systematic data to inform policy discussions and clinical care practice.

DETAILED DESCRIPTION:
Kidney transplantation extends and improves the lives of adults with end-stage renal disease (ESRD). Live donor kidney transplantation (LDKT) has many advantages over deceased donor transplantation for the recipient, including shorter or no dialysis exposure, immediate graft function, lower perioperative morbidity and mortality, and better long-term graft and patient survival. Also, it yields significant cost savings to the healthcare system overall. These relative advantages and other advances in the field (e.g., laparoscopic techniques, paired kidney exchanges) have led transplant candidates and programs to more proactively embrace LDKT as the primary treatment option. Living kidney donors now account for 40% of all kidney transplants performed in the United States during the past 10 years, and more than 90,000 adults have undergone living donor nephrectomy in the United States over the last 20 years.

Worldwide there have been few large-scale studies examining the short- and long-term outcomes of living kidney donation, and many have been limited by retrospective, cross-sectional, and/or single-center designs with no appropriate control group. Despite efforts to enhance understanding of donor outcomes, it is clear that we have more knowledge in some areas (e.g., surgical and short-term medical complications) than in others (e.g., long-term medical complications, psychological outcomes, financial impact). The relative paucity of multisite, prospective outcome studies is concerning, especially considering the expanding donor eligibility criteria used by transplant programs today. Over the past decade, criteria for acceptance of a living donor candidate has changed: some donor candidates who would not have been considered 15 years ago (e.g., those with hypertension, obesity, or no prior relationship with the recipient) are now readily evaluated by many programs.

Recently, the transplant community and changes in federal regulations have brought attention to the need for more systematic study of living donor outcomes. While reporting outcomes over a 2-yr period is now mandated by the Organ Procurement and Transplantation Network (OPTN) and the United Network for Organ Sharing (UNOS), most transplant programs do not systematically collect donor outcome data. The lack of such data is an important problem because, without it, we will continue to have considerable variability in informed consent processes for living donors and their recipients, as well as limited data to inform clinical practice and policy development. This study directly addresses several of the recommendations made by the U.S. Department of Health and Human Services' Advisory Committee on Organ Transplantation.

A. Design Overview

This is a six center, prospective observational cohort study. A total of 280 living kidney donors, 280 LDKT recipients, and 160 healthy comparison subjects meeting all eligibility criteria will be enrolled. Participants will complete the assessment protocol at 5 time points: prior to surgery (Baseline, T1), 1 month after surgery (T2), 6 months after surgery (T3), 12 months after surgery (T4), and 24 months after surgery (T5). The rationale for selecting these time points is that they correspond to the assessment intervals currently required by the OPTN/UNOS for living donor follow-up, which were selected by the Living Donation Committee as the most appropriate time points for gathering short- and long-term follow-up data.

B. Study Participants

A total of 280 living kidney donors, 280 LDKT recipients, and 160 healthy comparison subjects meeting all eligibility criteria will be enrolled.

We will enroll both English and Spanish speaking participants into the study. All questionnaire outcomes will be translated into Spanish using conventional translational procedures and we will ensure that an interviewer at BIDMC is fluent in Spanish. It is important to emphasize that not all of the questionnaires used in this study have been validated in Spanish or with Hispanic patients. While this is an important limitation, we feel that this limitation is outweighed by the potential benefits of including primarily Spanish-speaking participants in the study.

The primary focus of the study is on assessing donor outcomes. The rationale for including the recipient is to examine the role that recipient factors play in predicting donor outcomes. There is preliminary evidence that some aspects of the recipient's functioning (e.g., graft survival, QOL) are associated with certain functional and psychological outcomes in living donors.7,8,88 The inclusion of transplant recipients in the study permits further examination of this association over time and allows us to include other recipient variables that heretofore have been neglected (e.g., perceptions of the donor-recipient relationship). Also, we will recruit a healthy, non-donor comparison group. A healthy comparison group allows us to address the question, "What if I had not donated my kidney?" - a question that is often considered by donors. These will be adults who completed one or more parts of the donor evaluation, but who did not proceed further for various reasons (although none of them medical).

C. Participant Recruitment and Retention

The first participant will be enrolled into the study in September 2011. Recruitment time is scheduled for 24 months. The last study assessment, therefore, will be completed in August 2015. Target recruitment for each site is 47 donor-recipient pairs and 27 healthy comparisons.

Importantly, we will recruit living donors into the study regardless of their recipient's participation status. Even in the absence of the recipient's participation, we will obtain valuable data about donor outcomes. However, because this is first-and-foremost a study evaluating donor outcomes, if a donor does not consent to participate in the study, we will not approach their recipient about study participation.

Non-directed donors will be recruited into the study. If it's an anonymous donation, their recipient will not be approached about the study. In the case, only the donor will be enrolled. If the non-directed donor has established a relationship (albeit a new one) with the intended recipient, then we will attempt to enroll both the donor and the recipient into the study, just like any other donor-recipient pair.

Donors participating in a paired kidney donation program (KPD) will be recruited into the study. In this instance, we will enroll KPD donors and their intended recipient (i.e., the recipient with whom they are incompatible, not the recipient of their specific kidney).

For each transplant recipient enrolled in the study, we will determine if s/he had other potential donors who were initially screened or evaluated but who did not progress to donation surgery. This initial screening or evaluation may include an initial health history, ABO testing, and/or other preliminary tests. To qualify as a control subject, the non-donor may or may not have completed the entire evaluation, but none of the studies performed will have excluded them from donation. If an enrolled donor has more than one potential health control subject, we will attempt to recruit them all into the study.

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years old
* residential or cell phone service
* written informed consent
* medically cleared for donor nephrectomy (donor)
* medically cleared for transplant surgery (recipient)
* did not progress to donation, although medically eligible (control)
* completed preliminary labs (control)

Exclusion Criteria:

* inability or unwillingness to provide informed consent
* inability to speak and read English or Spanish

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A total of 280 living kidney donors, 280 LDKT recipients, and 160 healthy comparison subjects meeting all eligibility criteria will be enrolled.
  We will enroll both English and Spanish speaking participants into the study. All questionnaire outcomes will be translated into Spanish using conventional translational procedures and we will ensure that an interviewer at BIDMC is fluent in Spanish. It is important to emphasize that not all of the questionnaires used in this study have been validated in Spanish or with Hispanic patients. While this is an important limitation, we feel that this limitation is outweighed by the potential benefits of including primarily Spanish-speaking participants in the study.
Sampling Method: Non-Probability Sample
Enrollment: 720 (Estimated)
Dates: Start 2011-08; Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
Surgical Outcomes | 1, 6, 12, and 24 Months Post-Surgery
  Multiple surgical outcomes will be measured, including: operative time, surgical complications, re-operation, hospital length of stay, wound pain intensity, surgical scarring, and hospital readmissions.
Medical Outcomes | Baseline (pre-donation), 1, 6, 12, and 24 Months Post-Surgery
  Multiple medical outcomes will be measured, including: blood pressure, creatinine, body mass index, serum creatinine, 24 hr creatinine clearance, 24 hr protein, 24 hr albumin, fasting glucose, hemoglobin, total cholesterol, LDL, and HDL.
Functional Outcomes | Baseline, 1, 6, 12, and 24 Months Post-Surgery
  Several functional outcomes will be measured, including: health-related quality of life, fatigue, physical activity, and return to work/school.
Psychological Outcomes | Baseline, 1, 6, 12, and 24 Months Post-Surgery
  Multiple psychological outcomes will be measured, including: donation pressure/coercion, mood, body image, donation benefits, life satisfaction, fear of kidney failure, decision stability, and donor-recipient relationship.

SECONDARY OUTCOMES:
Costs | Baseline, 1, 6, 12, and 24 Months Post-Surgery
  We are assessing the financial impact of living kidney donation by assessing both direct and indirect costs associated with donor evaluation, surgical recovery and rehabilitation, and long-term recovery.

CONTACTS AND LOCATIONS:
Overall Officials: James R Rodrigue, Ph.D., Principal Investigator — Beth Israel Deaconess Medical Center; Didier Mandelbrot, M.D., Principal Investigator — Beth Israel Deaconess Medical Center
Locations (7):
- United States (7):
  - University of Arizona, Tucson, Arizona
  - University of Iowa, Iowa City, Iowa
  - Maine Medical Center, Portland, Maine
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Montefiore Medical Center, The Bronx, New York
  - Cleveland Clinic, Cleveland, Ohio
  - Rhode Island Hospital, Providence, Rhode Island

REFERENCES:
- [Derived] Rodrigue JR, Fleishman A, Sokas CM, Schold JD, Morrissey P, Whiting J, Vella J, Kayler LK, Katz D, Jones J, Kaplan B, Pavlakis M, Mandelbrot DA. Rates of Living Kidney Donor Follow-up: Findings From the KDOC Study. Transplantation. 2019 Jul;103(7):e209-e210. doi: 10.1097/TP.0000000000002721. No abstract available. PMID 31241558
- See also: Related Info — http://www.kdocstudy.com